CLINICAL TRIAL: NCT07290777
Title: A Phase 2, Randomized, Partially Blinded, Controlled, Dose-ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of VEL-101 in Kidney Transplant Recipients.
Brief Title: VEL-101 to Prevent Rejection After Kidney Transplantation
Acronym: RENGEVITY-201
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VEL-101.KI201
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Transplantation, Kidney
Keywords: Kidney transplant; VEL-101; pegrizeprument; renal allograft rejection; prophylaxis; kidney; renal; transplant; CD28 inhibitor; monoclonal antibody fragment; FR-104; Anti-CD28
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigator/participant blinded to VEL-101 dose level but not blinded to participants receiving tacrolimus.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VEL-101 Low Dose (Experimental): VEL-101 Low Dose
  Interventions: Drug: VEL-101
- VEL-101 High Dose (Experimental): VEL-101 High Dose
  Interventions: Drug: VEL-101
- Tacrolimus (Active Comparator): Tacrolimus
  Interventions: Drug: Tacrolimus (TAC)

INTERVENTIONS:
Drug: Tacrolimus (TAC) — Tacrolimus Immediate Release in addition to SOC
  Arms: Tacrolimus
Drug: VEL-101 — VEL-101 in addition to SOC
  Other Names: Pegrizeprument; FR104
  Arms: VEL-101 High Dose; VEL-101 Low Dose

SUMMARY:
This study will evaluate the safety and efficacy of VEL-101 compared with tacrolimus in patients undergoing kidney transplantation.

DETAILED DESCRIPTION:
This study is a randomized, multicenter, partially blinded, active control study to evaluate the safety and effectiveness of VEL-101 compared with tacrolimus in the prevention of rejection in patients undergoing kidney transplantation. Up to 120 de novo kidney transplant recipients will receive rATG with corticosteroids (CS), and mycophenolate as maintenance therapy, and will be randomized 1:1:1 to receive either VEL-101 (low dose or high dose) or tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age
2. Able to understand key components of the study as described in the written informed consent document and willing and able to provide written informed consent.
3. If female, surgically sterile (post hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), postmenopausal (greater than 12 months of amenorrhea without alternative medical causes), or, if of childbearing potential, is using a highly effective contraception until 90 days after EOS visit.
4. If male, is vasectomized, has undergone bilateral orchidectomy, agrees to abstinence of heterosexual intercourse, or only has female partner using highly effective contraception, surgically sterile or postmenopausal and agrees to use method until 90 days after EOS visit.
5. Receiving kidney allograft from deceased donor or non-human leukocyte antigen (HLA) identical living donor.

   a) Repeat kidney transplant allowed if no previous kidney transplant(s) failed due to recurrent disease within first year, acute rejection or nonsurgical thrombosis
6. Able & willing to comply with all study procedures, including PK and PD assessments, as assessed by the Investigator
7. Vaccination up to date per the center's SOC as assessed by the Investigator.
8. In the opinion of the Investigator, is able to adhere to the study requirements.

Exclusion Criteria:

1. Negative for EBV or Epstein-Barr nuclear antigen antibody
2. Know allergy to study medication (rATG, corticosteroids, MMF, tacrolimus, or VEL-101) or its components or a history of a severe allergic reaction to any drug.
3. History of previous non-kidney solid organ, vascular composite allograft, pancreatic islet, stem cell or bone marrow transplant.
4. Planned multiorgan transplant, including dual or en-bloc kidney transplant
5. Anticipated cold ischemia time (CIT) >30 hours
6. Donor with Kidney Donor Profile Index (KDPI) > 85%
7. Panel reactive antibody >80%, calculated panel-reactive antibody (CPRA)>80% or history of HLA desensitization
8. Positive T or B cell flow, cytotoxic, or virtual crossmatch at Screening
9. Current or historical DSA
10. Recipient or donor with positive hepatitis B surface antigen (HBsAG), hepatitis B core antibody (HBcAb), hepatitis B virus (HBV) nucleic acid testing (NAT), hepatitis C virus (HCV) antibody, HCV NAT, human immunodeficiency virus (HIV), or HIV NAT
11. Recipient who is CMV IgG negative (R-) receiving a kidney from a donor who is CMV IgG positive (D+)
12. Thrombocytopenia (platelets < 75,00/mm3), leukopenia (white blood cells [WBC] <3,000/mm3), or anemia (hemoglobin <8 g/dL) at Screening
13. History of inadequately treated active or latent mycobacterium tuberculosis (TB) infection
14. Clinically significant abnormality on 12-lead electrocardiogram (ECG) at Screening, as determined by the Investigator
15. Positive pregnancy test or lactating at Screening with plans to continue lactating regimen throughout the study
16. History of malignancy within the past 5 years (with the exception of non-metastatic basal or squamous cell carcinoma of the skin with successful treatment), or current active malignancy
17. Liver disease, defined as having elevated aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels greater than three times the upper value of the normal range of the study center at Screening
18. Medical condition requiring chronic use of daily prednisone doses >5 mg (or equivalent)
19. End-stage renal disease caused by primary focal segmental glomerulosclerosis (FSGS), atypical hemolytic uremic syndrome (aHUS), C3 glomerulopathy, or monoclonal gammopathy of kidney significance

    a) Note: participants with an unknown cause of ESRD can be included.
20. Participation in an investigational study within 30 days or within 5 half-lives of the investigational agent, whichever is longer, prior to Screening
21. Receiving any antibody or biologic medicinal product (with the exception of erythropoietin products) within 90 days prior to Screening
22. Positive test for SARS-CoV-2 antigen, polymerase chain reaction (PCR), or equivalent testing, at Screening, if performed
23. History or presence of coagulopathy, thrombophilia, unexplained bleeding or clotting disorders, or use of systemic anticoagulants at the time of transplant, with the exception of uremic coagulopathy or prophylactic heparin preparations.
24. History or presence, upon clinical evaluation, of any illness or condition that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the participant at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs) | Month 12
  Incidence of serious adverse events (SAEs)
Incidence of treatment emergent adverse events (TEAEs) | Month 12
  Incidence of treatment emergent adverse events (TEAEs)
PK Parameter Cmax | Day 1, Month 3
  PK Parameter Cmax
PK Parameter Cmin | Day 1, Month 3
  PK Parameter Cmin
PK Parameter Tmax | Day 1, Month 3
  PK Parameter Tmax
AUC from 0-8 hours | Day 1, Month 3
  AUC from 0-8 hours
AUC from 0 to 48 hours | Day 2
  AUC from 0 to 48 hours
VEL-101 Accumulation Ratio | Month 3
  VEL-101 Accumulation Ratio
VEL-101 Pre-Dose Serum Concentration | Day 1, Day 14, Months 1, 2, 3, 6, 9, 12, Periprocedural (kidney biospy)
  VEL-101 Pre-Dose Serum Concentration
Effect of Anti-Drug Antibody (ADA) Development on VEL-101 Serum Concentration | Months 1, 2, 3, 6, 9, 12, Periprocedural (kidney biopsy)
  Effect of Anti-Drug Antibody (ADA) Development on VEL-101 Serum Concentration
Effect of Neutralizing Antibody (NAb) Development on VEL-101 Serum Concentration | Day 1, Months 1, 2, 3, 6, 9, 12 and Periprocedural (kidney biopsy)
  Effect of Neutralizing Antibody (NAb) Development on VEL-101 Serum Concentration
VEL-101 CD28 Receptor Occupancy Concentration (%) | Days 1, 2, 3, 4, 5, 7, 14, 42, 70, 82, 91, 98 and Months 1, 2, 3, 6, 9, 12 and Periprocedural (kidney biopsy)
  VEL-101 CD28 Receptor Occupancy Concentration (%)

SECONDARY OUTCOMES:
Percentage Participants Meeting Composite Endpoint | Month 12
  Death, graft failure or biopsy proven acute rejection (BPAR, T cell mediated rejection [TCMR] Banff Grade > or = to 1A or antibody-mediated rejection [AMR] )
Slope of estimated glomerular filtration rage (eGFR) | Month 12
  Slope of estimated glomerular filtration rage (eGFR)
Incidence Injection Site Reaction | Month 12
  Incidence Injection Site Reaction
Incidence Adverse Events of Special Interest (AESIs) | Month 12
  AESIs Including BK viremia, BK virus-associate nephropathy, EBV viremia, PTLD, CMV viremia, CMV disease, malignancies
Proportion of Participants Discontinuing due to Adverse Events | Month 12
  Proportion of Participants Discontinuing due to Adverse Events
Incidence Delayed Graft Function Delayed Graft Function | Day 28
  Incidence Delayed Graft Function
Duration Delayed Graft Function | Day 28
  Duration Delayed Graft Function
Incidence of Renal Replacement Therapy (RRT) | Month 12
  Incidence of Renal Replacement Therapy (RRT)
Duration of Renal Replacement Therapy (RRT) | Month 12
  Duration of Renal Replacement Therapy (RRT)
Incidence of New-Onset Diabetes after Transplantation (NODAT) | Month 12
  Incidence of New-Onset Diabetes after Transplantation (NODAT)
Effect of Anti-Drug Antibody (ADA) Formation on VEL-101 t1/2 (hours) | Months 1, 2, 3, 6, 9, 12 and Periprocedural (kidney biopsy)
  Effect of Anti-Drug Antibody (ADA) Formation on VEL-101 t1/2 (hours)
Effect of Anti-Drug Antibody (ADA) Development on VEL-101 Volume of distribution (liters) | Months 1, 2, 3, 6, 9, 12 and Periprocedural (kidney biopsy)
  Effect of Anti-Drug Antibody (ADA) Development on VEL-101 Volume of distribution (liters)
Effect of Anti-Drug Antibody Development on VEL-101 Cmin (ng/mL) | Months 1, 2, 3, 6, 9, 12 and Periprocedural (kidney biopsy)
  Effect of Anti-Drug Antibody Development on VEL-101 Cmin (ng/mL)
Effect of Anti-Drug Antibody Development on VEL-101 Cmax (ng/mL) | Months 1, 2, 3, 6, 9, 12 and Periprocedural (kidney biopsy)
  Effect of Anti-Drug Antibody Development on VEL-101 Cmax (ng/mL)

IPD SHARING:
Plan to Share IPD: No